CLINICAL TRIAL: NCT05826327
Title: Effects of Epidural Labor Analgesia With Esketamine on the Incidence of Postpartum Depression and Maternal and Neonatal Outcomes in Parturients With Prenatal Depression
Brief Title: Effects of Epidural Labor Analgesia With Esketamine on the Incidence of Postpartum Depression in Parturients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Peking University First Hospital (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); Beijing Obstetrics and Gynecology Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-20230021-R
Record Dates: First submitted 2023-03-19; First posted 2023-04-24 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-05

CONDITIONS: Postpartum Depression
Keywords: Esketamine; Epidural labor analgesia; Postpartum depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Esketamine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Esketamine Group (Experimental): The epidural analgesic drug mix for labour analgesia is ropivacaine 0.08mg/mL compounded with esketamine 0.3mg/mL.
  Interventions: Drug: Esketamine
- Control Group (Placebo Comparator): The epidural analgesic drug mix for labour analgesia is ropivacaine 0.08mg/mL compounded with sufentanil 0.3ug/mL.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Esketamine — The drug esketamine will be added to the experimental group as opposed to the control group.
  Other Names: E
  Arms: Esketamine Group
Drug: Sufentanil — Sufentanil for labour analgesia in the control group
  Other Names: C
  Arms: Control Group

SUMMARY:
Postpartum depression is a common psychological abnormality during the puerperium, which seriously affects maternal and neonatal health. Esketamine, the S-enantiomer of ketamine, is twice as potent as ketamine and can be safely used for cesarean section and labor analgesia. However, it is not clear whether esketamine used for epidural labor analgesia can significantly reduce the incidence of postpartum depression. This study intends to explore the incidence of maternal prenatal depression and to investigate the effect of esketamine for epidural labor analgesia on postpartum depression and maternal and neonatal outcomes in parturients with prenatal depression through a multi-center, large-scale and high-quality clinical trail, in order to provide a clinical basis and theoretical basis for the application of esketamine used for epidural labor analgesia in postpartum depression and further reduce the incidence of postpartum depression, promote maternal and infant health, and ensure maternal and infant safety .

DETAILED DESCRIPTION:
The study include women who meet the inclusion criteria for antenatal EPDS score ≥10 for labour analgesia while signing informed consent. The women will be randomized into two groups, one for esketamine group and the other for the control group. Follow-up visits will be conducted at 1 day, 7 days and 42 days after delivery. The primary endpoint of the study was the incidence (MINI-6.0 for diagnosis of postnatal depression) and severity of maternal depression at day 42 postpartum. The secondary endpoints of the study are maternal EPDS scores at 7 and 42 days postpartum; pain scores and impact at 1, 7 and 42 days postpartum; breastfeeding at 1, 7 and 42 days postpartum; length of postpartum stay; maternal complications at 42 days postpartum and neonatal illnesses at 42 days postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Full-term pregnancy; Antenatal depressive state (EPDS score ≥10 and non-depressive diagnosis by a psychiatrist); Epidural labor analgesia； Signed informed consent.

Exclusion Criteria:

* Pre-existing history of definite psychiatric disorders (depression, schizophrenia, etc.) or communication disorders；Presence of severe preoperative pregnancy complications (e.g., severe preeclampsia, placental implantation, HELLP syndrome, placenta praevia, placenta abruptio)；ASA classification ≥ grade III；Contraindications to ketamine/S-ketamine (e.g., intractable, refractory hypertension, severe cardiovascular disease [cardiac function class ≥ III], hyperthyroidism); Refusal to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of depression | Day 42 after completion of labour
  The incidence (MINI-6.0 for the diagnosis of postnatal depression) and severity of depression on day 42 after delivery in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Lyv, Dr, Study Director — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's hospital, school of medicine, Zhejiang university, Hangzhou, Zhejiang, China